CLINICAL TRIAL: NCT02744131
Title: OCP vs Metformin for Improvement in Clinical Symptoms and Metabolic Markers in Indian PCOS Women
Acronym: OCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kar Clinic & Hospital Pvt. Ltd. (Other)
Collaborators: All India Institute of Medical Sciences (Other); Nova IVI Fertility, New Delhi (Unknown); Dr Patil's Fertility & Endoscopy Clinic, Bangalore (Unknown); Shreyas Hospital & Sushrut Assisted Conception Clinic, Kolhapur (Unknown); University of Messina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCP-MET-2016
Record Dates: First submitted 2016-03-20; First posted 2016-04-20 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; Metformin; OCP; metabolic parameters
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Contraceptives, Oral; Cyproterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCP (Active Comparator): Arm 1: oral contraceptive pill, combination pill of ethyl estradiol 20 micro gram with Cyproterone acetate.
  Interventions: Drug: Oral contraceptive pill combination of ethyl estradiol and Cyproterone acetate
- Metformin (Active Comparator): Arm 2: Metformin . Oral insulin sensitising drug in the dose of 1500gms daily.
  Interventions: Drug: Metformin 1500mgs per day

INTERVENTIONS:
Drug: Oral contraceptive pill combination of ethyl estradiol and Cyproterone acetate
  Arms: OCP
Drug: Metformin 1500mgs per day
  Arms: Metformin

SUMMARY:
Objective: To assess effectiveness of ISD (Insulin sensitizing drugs) Vs OCP (Combined E&P cyproterone acetate) in improving clinical, hormonal and metabolic features of PCOS( polycystic ovary syndrome)women from India.

Intervention:

Randomized to receive Metformin 1500 mg / day OR OCP (EE+CA) Life style advice to women with BMI ( body mass index) more than 28 , in both groups (PS: progesterone can be added for getting withdrawal bleeding for amenorrhoea of more than two months, or for prolonged menstrual bleeding. ) Study period: 6 months Clinical evaluation points and tests at enrollment and again after 6 month. Clinical: BMI, Waist circumference, Hip circumference, Acne score, FG (modified Ferriman Gallwey score ) (after no epilation for last 6 weeks), Menstrual History Biochemical: Thyroid function tests, Prolactin,Total Testosterone, Lipid Profile, FAsting blood sugar & 75 gm 2 hr Glucose tolerance test (GTT), Sr Insulin, 25- hydroxy vitamin D (optional), (Only Radioimmunoassay / Chemiluminescence assays)

Acronyms: OCP(oral contraceptive pills); PCOS (polycystic ovary syndrome); FBS(fasting blood sugar); GTT(glucose tolerance test)

ELIGIBILITY:
Inclusion Criteria:

* PCOS Women diagnosed by Rotterdam criteria
* Age > 16 or menarche of at least 2 yr upto age 40.
* Diagnosed by Rotterdam Anovulation F.G. Score ≥ 8 or Total testosterone ≥ 40 ngms/dl ovarian volume ≥ 10 cc BMI>23
* Women not attempting pregnancy at present.

Exclusion Criteria:

* PCOS Women with BMI ≤ 23
* Undergoing any treatment for acne hirsutism. Including Homeopathic, Ayurvedic
* Known diabetic or hypertension .

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Improvements in Menstrual cycle in women with polycystic ovary syndrome. | Six months
  To compare improvement in Menstrual cycle. Women will be required to maintain a menstrual calendar for the duration of the study and asked to fill a questionnaire before and after study duration.The questionnaire will cover menstrual cycle dates, duration and amount. Interpreting the answered will help in assessing improvement in menstrual pattern.
Improvement in hirsutism | six months
  FG scores before and after treatment will be compared between the two arms. Modified Ferriman and Gallwey visual score will be used by a nurse to assess before and after the study period.
Improvement in acne score | Six months
  Acne scores before and after treatment will be compared between the two arms. Visual assessment of acne using "mild/moderate/severe " grades will be assessed before and after study by a physician.
Weight loss following treatment | 6months
  Weight loss will be compared between the two arms following 6 months of treatment
Reduction in total testosterones | 6months
  Reduction in total testosterones, signifying biochemical hyperandrogenemia, will be compared between the two groups following 6 months treatment.
Reduction in serum fasting insulin | 6 months
  Reduction in insulin levels following treatment will be compared between the two arms
Improvements in lipid profile | 6months
  Any improvement in triglycerides and HDLc (high density lipoprotein c) will be compared between the two groups after 6 months of treatment
Improvement in glucose tolerance | 6months
  75grams 2 hour glucose challenge test results will be compared pre and post treatment between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- KAR clinic and hospital pvt ltd, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kar S. Clomiphene citrate or letrozole as first-line ovulation induction drug in infertile PCOS women: A prospective randomized trial. J Hum Reprod Sci. 2012 Sep;5(3):262-5. doi: 10.4103/0974-1208.106338. PMID 23531705
- [Background] Kar S, Sanchita S. Clomiphene citrate, metformin or a combination of both as the first line ovulation induction drug for Asian Indian women with polycystic ovarian syndrome: A randomized controlled trial. J Hum Reprod Sci. 2015 Oct-Dec;8(4):197-201. doi: 10.4103/0974-1208.170373. PMID 26752854
- [Background] Kumar P, Nawani N, Malhotra N, Malhotra J, Patil M, Jayakrishnan K, Kar S, Jirge PR, Mahajan N. Assisted reproduction in polycystic ovarian disease: A multicentric trial in India. J Hum Reprod Sci. 2013 Jan;6(1):49-53. doi: 10.4103/0974-1208.112382. PMID 23869152